CLINICAL TRIAL: NCT01877083
Title: A Multicenter, Open-Label, Phase 2 Study of the Safety and Activity of Lenvatinib (E7080) in Subjects With KIF5B-RET-Positive Adenocarcinoma of the Lung
Brief Title: Study of the Safety and Activity of Lenvatinib (E7080) in Subjects With KIF5B-RET-Positive Adenocarcinoma of the Lung
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7080-G000-209
Record Dates: First submitted 2013-06-11; First posted 2013-06-13 (Estimated); Results first posted 2019-08-13 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2018-01

CONDITIONS: KIF5B-RET-Positive Adenocarcinoma of the Lung
Keywords: KIF5B-RET-Positive Adenocarcinoma; Lung Cancer; NSCLC; Non-Small Cell Lung Cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lenvatinib (Experimental)
  Interventions: Drug: Lenvatinib

INTERVENTIONS:
Drug: Lenvatinib — Starting dose of 24 mg orally, once per day
  Other Names: E7080

SUMMARY:
This is a Phase 2, open-label, safety and activity study of lenvatinib in subjects with KIF5B-RET-positive adenocarcinoma of the lung and other confirmed RET translocations. At least 20 subjects with KIF5B-RET and other RET translocations will be treated and will receive lenvatinib at a starting dose of 24 mg orally, once per day. The study will consist of 3 phases: The Pretreatment Phase, The Treatment Phase and the Extension Phase. The Pretreatment Phase will include screening procedures and eligibility assessments. The Pretreatment Phase consists of a Screen 1, Screen 2 and Baseline Period. The Treatment Phase will begin when the subject has met all eligibility criteria on Day 1 of the first Treatment Cycle. The Treatment Phase contains the Treatment and Follow-up Periods. The Extension Phase will begin for subjects who received treatment in the study (either in the Treatment Period or Follow-up Period) at the time of database cutoff.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have a cytological or histological confirmed diagnosis of adenocarcinoma of the lung.
2. Subject must be known to be RET positive (known KIF5B-RET translocation, or other confirmed RET translocations (e.g., CCDC6-RET)) or have an available tumor sample for local or central testing obtained prior to consent (Screen 1). Subjects whose samples need to be submitted for central laboratory testing must be current non-smokers and not known to have mutation in EGFR, KRAS, or ALK.
3. Subjects may have received up to three prior systemic anticancer treatment regimens for adenocarcinoma of the lung (including adjuvant therapies and tyrosine-kinase inhibitors [TKI]), unless discussed with the sponsor.
4. Subjects must have a clinically indicated need for systemic chemotherapy for adenocarcinoma of the lung based on the investigator's assessment
5. Presence of measurable disease meeting the following criteria:

   1. At least one lesion of at least 1.0 cm in the long-axis diameter for a non-lymph node or at least 1.5 cm in the short-axis diameter for a lymph node which is serially measurable according to Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) using either computerized tomography (CT) or magnetic resonance imaging (MRI). If there is only one target lesion and it is a non-lymph node, it should have a longest diameter of at least 1.5 cm.
   2. Lesions previously treated with radiotherapy or locoregional therapy must show radiographic evidence of disease progression to be deemed a target lesion.
6. Subjects with known brain metastases who have completed whole brain radiotherapy, stereotactic radiosurgery, or complete surgical resection will be eligible if they have remained clinically stable, asymptomatic and off of steroids for 28 days.
7. Adequate bone marrow function, defined as:

   1. Absolute neutrophil count (ANC) greater than or equal to 1.5 x 10^9/L (greater than or equal to 1500/mm^3)
   2. Hemoglobin (Hb) greater than or equal 8.5 g/dL
   3. Platelet count greater than or equal 75 x 10^9/L (greater than or equal 75,000/mm^3)
8. Adequate liver function, defined as:

   1. Bilirubin less than or equal 1.5 x upper limit of normal (ULN) except for unconjugated hyperbilirubinemia or Gilbert's syndrome
   2. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase (ALP) less than or equal 3 x ULN (less than or equal 5 x ULN if subject has liver metastases). If alkaline phosphatase is greater than 3 x ULN (in absence of liver metastases) or greater than 5 x ULN (in presence of liver metastases) AND the subject also is known to have bone metastases, the liver-specific alkaline phosphatase must be separated from the total and used to assess the liver function instead of total alkaline phosphatase.
9. Adequate renal function, defined as calculated creatinine clearance greater than 40 mL/min per the Cockcroft and Gault formula.
10. Adequately controlled blood pressure (BP) with or without antihypertensive medications, defined as BP less than 150/90 mmHg at screening and no change in antihypertensive medications within 1 week before Cycle 1/Day 1 (C1D1).
11. Eastern Cooperative Oncology Group (ECOG)-Performance Status (PS) of 0 or 1.
12. Survival expectation of 12 weeks or longer after starting study drug.
13. Males or females aged at least 18 years (or any age greater than 18 years as determined by country legislation) at the time of informed consent (Screen 1).
14. Females must not be breast-feeding or pregnant at Screening or Baseline (as documented by a negative beta-human chorionic gonadotropin [B-hCG] test with a minimum sensitivity of 25 IU/L or equivalent units of B-hCG). A separate baseline assessment is required if a negative Screening pregnancy test was obtained more than 72 hours before the first dose of study drug.
15. All females will be considered to be of childbearing potential unless they are postmenopausal (amenorrheic for at least 12 consecutive months, in the appropriate age group and without other known or suspected cause) or have been sterilized surgically (i.e., bilateral tubal ligation, total hysterectomy or bilateral oophorectomy, all with surgery at least one month before dosing).
16. Females of childbearing potential must not have had unprotected sexual intercourse within 30 days before study entry and must agree to use a highly effective method of contraception (e.g., total abstinence, an intrauterine device, a double-barrier method [such as condom plus diaphragm with spermicide], a contraceptive implant, an oral contraceptive, or have a vasectomized partner with confirmed azoospermia) throughout the entire study period and for 30 days after study drug discontinuation. If currently abstinent, the subject must agree to use a double barrier method as described above if she becomes sexually active during the study period or for 30 days after study drug discontinuation. Females who are using hormonal contraceptives must have been on a stable dose of the same hormonal contraceptive product for at least 4 weeks before dosing and must continue to use the same contraceptive during the study and for 30 days after study drug discontinuation.
17. Male subjects must have had a successful vasectomy (confirmed azoospermia) or they and their female partners must meet the criteria above (i.e., not of childbearing potential or practicing highly effective contraception throughout the study period and for 30 days after study drug discontinuation). No sperm donation is allowed during the study period and for 30 days after study drug discontinuation.
18. Provide written informed consent (Screen 1 and Screen 2)
19. Willing and able to comply with all aspects of the protocol

Exclusion Criteria:

1. Subjects who have received any anticancer therapy (including surgery, locoregional, biological, immunotherapy, hormonal, or radiotherapy) within 21 days before the first dose of study drug (28 days for investigational therapies).
2. Leptomeningeal metastases or brain metastases except as for Inclusion Criterion #6.
3. Subjects who have not recovered from toxicities as a result of prior anticancer therapy to less than Grade 2 severity per the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v4.0, except alopecia and infertility.
4. Significant cardiovascular impairment: history of congestive heart failure greater than New York Heart Association (NYHA) Class II, unstable angina, myocardial infarction, or stroke within 6 months of the first dose of study drug, or cardiac arrhythmia requiring medical treatment at Screening.
5. Gastrointestinal malabsorption or any other condition in the opinion of the investigator that might affect the absorption of lenvatinib.
6. Active malignancy (except for adenocarcinoma of the lung or definitively treated melanoma in-situ, basal or squamous cell carcinoma of the skin, or carcinoma in-situ of the cervix) within the past 24months.
7. Major surgery within 3 weeks before the first dose of study drug.
8. Bleeding or thrombotic disorders or use of anticoagulants such as warfarin or similar agents requiring therapeutic international normalized ratio (INR) monitoring. (Treatment with low molecular weight heparin is allowed.)
9. Active hemoptysis (bright red blood of at least 0.5 teaspoon) within 3 weeks before the first dose of study drug.
10. Active infection (any infection requiring treatment).
11. Symptomatic central nervous system (CNS) disease.
12. Subjects having greater than 1+ proteinuria on urine dipstick testing will undergo 24-hour urine collection for quantitative assessment of proteinuria. Subjects with urine protein greater than or equal to 1 g/24-hour will be ineligible.
13. Any medical or other condition that in the opinion of the investigator(s) would preclude the subject's participation in a clinical study or would preclude them from completing the study.
14. Scheduled for surgery during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-04-05 (Actual); Primary Completion 2016-02-03 (Actual); Study Completion 2017-11-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (23):
- United States (8):
  - Duarte, California
  - La Jolla, California
  - Whittier, California
  - Jacksonville, Florida
  - Canton, Ohio
  - Cleveland, Ohio
  - Knoxville, Tennessee
  - Dallas, Texas
- Hong Kong (2):
  - Hong Kong
  - Shatin
- Japan (9):
  - Nagoya, Aichi-ken
  - Kashiwa, Chiba
  - Akashi, Hyōgo
  - Kobe, Hyōgo
  - Natori-shi, Miyagi
  - Ōsaka-sayama, Osaka
  - Chuo-ku, Tokyo
  - Koto-Ku, Tokyo
  - Fukuoka
- Singapore (2):
  - National Cancer Center Hospital, Singapore
  - National University Hospital, Singapore
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Veterans General Hospital Taipei, Taipei

REFERENCES:
- [Derived] Hida T, Velcheti V, Reckamp KL, Nokihara H, Sachdev P, Kubota T, Nakada T, Dutcus CE, Ren M, Tamura T. A phase 2 study of lenvatinib in patients with RET fusion-positive lung adenocarcinoma. Lung Cancer. 2019 Dec;138:124-130. doi: 10.1016/j.lungcan.2019.09.011. Epub 2019 Sep 16. PMID 31710864
- [Derived] Wu H, Shih JY, Yang JC. Rapid Response to Sunitinib in a Patient with Lung Adenocarcinoma Harboring KIF5B-RET Fusion Gene. J Thorac Oncol. 2015 Sep;10(9):e95-e96. doi: 10.1097/JTO.0000000000000611. No abstract available. PMID 26291023

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 14 investigative sites in the United States, Japan, Singapore, and Taiwan from 05 April 2013 to 2 November 2017.
Pre-assignment Details: A total of 25 participants with kinesin family 5B oncogene rearranged during transfection (KIF5B-RET)-positive adenocarcinoma of the lung or other RET translocations were enrolled and treated, 5 participants were ongoing in the Extension Phase at the time of data cut-off.
Groups:
- Lenvatinib 24 mg: Participants with KIF5B-RET-positive adenocarcinoma and other RET translocations received lenvatinib 24 milligram (mg), capsule, orally, once daily in 28-day continuous cycles until disease progression (PD), development of unacceptable toxicity, withdrawal of consent, or termination of lenvatinib development by the sponsor.
Period: Treatment Phase
Arm/Group | Lenvatinib 24 mg
Started | 25
Completed | 5
Not Completed | 20
Not completed — Disease Progression | 10
Not completed — Clinical Progression | 1
Not completed — Adverse Event | 6
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 1
Period: Extension Phase
Arm/Group | Lenvatinib 24 mg
Started | 5
Completed | 0
Not Completed | 5
Not completed — Disease Progression | 3
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all participants who received at least 1 dose of lenvatinib.
Groups:
- Lenvatinib 24 mg: Participants with KIF5B-RET-positive adenocarcinoma and other RET translocations received lenvatinib 24 mg, capsule, orally, once daily in 28-day continuous cycles until PD, development of unacceptable toxicity, withdrawal of consent, or termination of lenvatinib development by the sponsor.
Arm/Group | Lenvatinib 24 mg
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.0 (13.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 17
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants with a best overall response (BOR) of complete response (CR) or partial response (PR), based on the investigator assessment of radiologic response according to Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1. No independent review of tumor assessments was performed. CR was defined as disappearance of all target lesions. Any pathological lymph nodes (target or non-target) had to be reduced in short axis to less than (<) 10 millimeter (mm). PR was defined as at least a 30% decrease in sum of diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: From first dose date until PD, development of unacceptable toxicity, withdrawal of consent, participant's choice to stop study treatment (up to approximately 2 years 10 months)
Population: FAS included all participants who received at least 1 dose of lenvatinib.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lenvatinib 24 mg
Number analyzed (Participants) | 25
percentage of participants | 16.0 [4.5 to 36.1]

2. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from the first dose to the date of first documentation of PD, or date of death, whichever occurred first. Tumor response data used to analyze PFS was obtained from the investigator's assessment of the imaging scans using RECIST 1.1. No independent review of tumor assessments were performed. PFS was calculated using Kaplan-Meier estimate and presented with 2-sided 95% Cl based on the Greenwood formula. PD was defined as at least 20% increase (including an absolute increase of at least 5 mm) in the sum of diameters of target lesions.
Time Frame: From first dose date until PD or death (up to approximately 2 years 10 months)
Population: FAS included all participants who received at least 1 dose of lenvatinib.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenvatinib 24 mg
Number analyzed (Participants) | 23
months | 7.3 [3.6 to 10.2]

3. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of first dose to the date of death from any cause. OS was calculated using Kaplan-Meier estimate and presented with 2-sided 95% Cl based on the Greenwood formula.
Time Frame: From first dose date until date of death from any cause (approximately up to 2 years 10 months)
Population: FAS included all participants who received at least 1 dose of lenvatinib.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenvatinib 24 mg
Number analyzed (Participants) | 25
months | NA [5.8 to NA] — Median and upper limit of confidence interval could not be calculated because higher number of participants were censored from analysis.

4. Secondary Outcome: Plasma Concentrations of Lenvatinib
Time Frame: Cycle 1 Day 1: 0.5-4 hours, 6-10 hours postdose; Cycle 1 Day 15: predose, 0.5-4 hours, 6-10 hours postdose; Cycle 2 Day 1: predose, 2-12 hours postdose; Cycle 3 Day 1: predose; (Cycle length is equal to [=] 28 days)
Population: The pharmacokinetic (PK) Analysis Set included all participants who received at least one dose of lenvatinib and had at least one quantifiable lenvatinib concentration. Participants who were evaluable at a particular time point for this outcome measure were included in the assessment.
Measure: Median (Full Range); unit: microgram per milliliter (mcg/mL)
Arm/Group | Lenvatinib 24 mg
Number analyzed (Participants) | 24
microgram per milliliter (mcg/mL)
  Cycle 1 Day 1: 0.5 to 4 hours postdose | 37.0 [NA to 529] — The lower range could not be calculated because concentration values were below level of quantification.
  Cycle 1 Day 1: 6 to 10 hours postdose | 278.5 [127 to 382]
  Cycle 1 Day 15: predose: number analyzed (Participants) | 21
  Cycle 1 Day 15: predose | 83.6 [31 to 201]
  Cycle 1 Day 15: 0.5 to 4 hours postdose: number analyzed (Participants) | 22
  Cycle 1 Day 15: 0.5 to 4 hours postdose | 89.2 [40 to 1390]
  Cycle 1 Day 15: 6 to 10 hours postdose: number analyzed (Participants) | 22
  Cycle 1 Day 15: 6 to 10 hours postdose | 277.5 [59 to 684]
  Cycle 2 Day 1: predose: number analyzed (Participants) | 17
  Cycle 2 Day 1: predose | 66.4 [21 to 272]
  Cycle 2 Day 1: 2 to 12 hours postdose: number analyzed (Participants) | 13
  Cycle 2 Day 1: 2 to 12 hours postdose | 345.0 [110 to 576]
  Cycle 3 Day 1: predose: number analyzed (Participants) | 13
  Cycle 3 Day 1: predose | 59.8 [27 to 522]

ADVERSE EVENTS:
Time Frame: From the first dose of study drug up to 30 days after the last dose of study drug (approximately up to 4 years 7 months)
Arm/Group | Lenvatinib 24 mg
All-Cause Mortality (participants affected / at risk) | 13/25
Serious Adverse Events (participants affected / at risk) | 16/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenvatinib 24 mg (N=25)
Cardiac failure (Cardiac disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Malaise (General disorders) | 1
Pyrexia (General disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Device related sepsis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 3
Transient ischaemic attack (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Bacterial infection (Infections and infestations) | 1
Ureteric stenosis (Renal and urinary disorders) | 1
Malignant pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lenvatinib 24 mg (N=25)
Anaemia (Blood and lymphatic system disorders) | 2
Hypothyroidism (Endocrine disorders) | 3
Dry eye (Eye disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 3
Abdominal pain upper (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 6
Diarrhoea (Gastrointestinal disorders) | 13
Dry mouth (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 14
Oral pain (Gastrointestinal disorders) | 2
Stomatitis (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 10
Fatigue (General disorders) | 9
Generalised oedema (General disorders) | 2
Malaise (General disorders) | 2
Oedema peripheral (General disorders) | 5
Pyrexia (General disorders) | 2
Pharyngitis (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 2
Alanine aminotransferase increased (Investigations) | 5
Aspartate aminotransferase increased (Investigations) | 6
Blood creatinine increased (Investigations) | 3
Neutrophil count decreased (Investigations) | 3
Platelet count decreased (Investigations) | 7
Weight decreased (Investigations) | 5
White blood cell count decreased (Investigations) | 2
Decreased appetite (Metabolism and nutrition disorders) | 13
Dehydration (Metabolism and nutrition disorders) | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Dysgeusia (Nervous system disorders) | 2
Headache (Nervous system disorders) | 10
Anxiety (Psychiatric disorders) | 2
Confusional state (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 2
Proteinuria (Renal and urinary disorders) | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 4
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 3
Hypertension (Vascular disorders) | 17
Hypotension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other